CLINICAL TRIAL: NCT05338853
Title: Comparative Effects of Gongs Mobilization and Scapular Mobilization on Pain, Range of Motion and Disability in Adhesive Capsulitis
Brief Title: Comparative Effects of Gongs Mobilization and Scapular Mobilization on Adhesive Capsulitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0103
Record Dates: First submitted 2022-04-15; First posted 2022-04-21 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive capsulitis, Gong's mobilization,
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gongs Mmobilization (Experimental): to deal adhesive capsulitis
  Interventions: Other: Gongs mobilization
- scapular mobilization (Experimental): to deal adhesive capsulitis
  Interventions: Other: scapular mobilization

INTERVENTIONS:
Other: Gongs mobilization — to deal adhesive capsulitis
  Arms: Gongs Mmobilization
Other: scapular mobilization — scapular mobilization
  Arms: scapular mobilization

SUMMARY:
Adhesive Capsulitis also known as frozen shoulder is a self-limiting disorder of the shoulder joint characterized by pain, loss of joint ROM and functional limitation which usually resolves in 12-15 months. I Different physical therapy techniques and modalities have been used in reducing pain and increasing ROM in frozen shoulder.

It is a randomized clinical trial and random sampling was used with an inclusion criterion of confirmed adhesive capsulitis patients. This study aims to provide a comparative analysis of two mobilizations: Gongs and Scapular mobilization in terms of effects on pain, range of motion and functional status. Patients having acute inflammation, fracture, dislocation or any surgery around the shoulder joint were excluded from the study. Subjects were randomly allocated into two groups with group A receiving Gongs mobilization and group B receiving scapular mobilization in addition to Continuous passive motion which was given as a baseline therapy to both the groups. Total duration of the study was 6 months. Numeric pain rating scale, universal goniometry and Shoulder pain and disability index were used to measure the pain, range of motion and functionality respectively at the start and end of study. After collecting data from defined study setting, data was entered and analyzed by using Statistical Package for the Social Sciences (SPSS) for Windows software, version 25. After assessing normality of data by Shapiro-Wilk test, it was decided either parametric or non-parametric test to be used.

DETAILED DESCRIPTION:
Adhesive Capsulitis also known as frozen shoulder is a self-limiting disorder of the shoulder joint characterized by pain, loss of joint ROM and functional limitation which usually resolves in 12-15 months. It develops when the glenohumeral capsule undergoes inflammation and is fibrosed as a result. Shoulder of an Adhesive capsulitis patient undergoes three stages; Freezing(0-6 months), Frozen (4 months-6 months) and Thawing(6 months- 2 years). Physical therapy is of considerable importance in management of adhesive capsulitis patients. Different physical therapy techniques and modalities have been used in reducing pain and increasing ROM in frozen shoulder.

It is a randomized clinical trial and random sampling was used with an inclusion criterion of confirmed adhesive capsulitis patients. This study aims to provide a comparative analysis of two mobilizations: Gongs and Scapular mobilization in terms of effects on pain, range of motion and functional status. Patients having acute inflammation, fracture, dislocation or any surgery around the shoulder joint were excluded from the study. Subjects were randomly allocated into two groups with group A receiving Gongs mobilization and group B receiving scapular mobilization in addition to Continuous passive motion which was given as a baseline therapy to both the groups. Total duration of the study was 6 months. Numeric pain rating scale, universal goniometry and Shoulder pain and disability index were used to measure the pain, range of motion and functionality respectively at the start and end of study. After collecting data from defined study setting, data was entered and analyzed by using Statistical Package for the Social Sciences (SPSS) for Windows software, version 25. After assessing normality of data by Shapiro-Wilk test, it was decided either parametric or non-parametric test to be used.

ELIGIBILITY:
Inclusion Criteria:

Confirmed Adhesive Capsulitis patients (Stage 2 and 3)

* ROM restriction in capsular pattern (External rotation > abduction > internal rotation)
* Functional tests positive (Hand to neck, hand to scapula)
* Both active and passive movement ranges limited.
* Males and Females of age 40-60 years

Exclusion Criteria:

1. Stage 1 Adhesive Capsulitis.
2. Acute inflammation
3. Recent fracture in and around the shoulder
4. Recent shoulder dislocation
5. Past surgery around shoulder joint

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 4months
  The 11-point NPRS consists of numbers between 0 and 10 where 0 indicates "no pain" and 10 indicates "maximum pain." The respondent is instructed to identify one number between 0 and 10, which is best representative of their pain intensity.
Degree of Range of motion | 4 months
  goniometer will be used to take ranges
The Shoulder Pain and Disability Index (SPADI) | 4 months
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rabiya Noor, PhD, Study Chair — Riphah International University
Locations (1):
- Railway Hospital, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No